CLINICAL TRIAL: NCT00781937
Title: Effect of Liraglutide on Long-term Weight Maintenance and Additional Weight Loss Induced by a 4 to 12 Week Low Calorie Diet in Obese Subjects; A 56 Week Randomised, Double-blind, Placebo Controlled, Parallel Group, Multicentre Trial With a 12 Week Follow-up Period
Brief Title: Comparison of Liraglutide Versus Placebo in Weight Loss Maintenance in Obese Subjects: SCALE - Maintenance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8022-1923
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2011-11-28 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lira 3.0 mg (Experimental): A 12-week run-in period where screened subjects were treated with a low calorie diet. Randomised subjects (those who lost more than or equal to 5% of screening body weight) were treated with liraglutide 3.0 mg, once daily, injected subcutaneously and instructed to follow a standard energy-restricted diet in the 56-week main trial period. Subjects discontinued treatment in the 12-week follow-up period. The starting dose of liraglutide was 0.6 mg, with weekly increments of 0.6 mg every 7 days until the target dose of 3.0 mg was reached
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator): A 12-week run-in period where screened subjects were treated with a low calorie diet. Randomised subjects (those who lost more than or equal to 5% of screening body weight) were treated with liraglutide placebo, once daily, injected subcutaneously for 56 weeks and instructed to follow a standard energy-restricted diet in the 56-week main trial period. Subjects discontinued treatment in the 12-week follow-up period
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Liraglutide 3.0 mg per day administered in a 6.0 mg/mL, 3 mL FlexPen® for subcutaneous (under the skin) injection, once daily
  Arms: Lira 3.0 mg
Drug: placebo — Liraglutide placebo 3 mL FlexPen® for subcutaneous (under the skin) injection, once daily
  Arms: Placebo

SUMMARY:
This trial is conducted in North America. The aim of this clinical trial is to evaluate the potential of liraglutide to maintain long term weight loss in obese non-diabetic subjects, as well as in overweight subjects who have medical problems such as hypertension (high blood pressure) or dyslipidaemia (an abnormal amount of lipids in the blood).

Trial has following trial periods: A 12-week run-in period (from week -12 to week 0) followed by a 56-week main trial period (weeks 0-56) and a 12-week follow-up period (weeks 56-68).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of either 30 kg/m^2 or more or BMI of less than 30 kg/m^2 to 27 kg/m^2 with presence of co-morbidities
* Stable body weight during the previous 3 months (less than 5 kg self-reported weight change)
* Previously undergone dietary weight loss and was not able to maintain reduced weight

Exclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes
* Previous treatment with GLP-1 (glucagon-like peptide-1) receptor agonists (including liraglutide or exenatide), within the last 3 months
* Visit 1 thryoid stimulating hormone (TSH) outside of the range of 0.4-6.0 mIU/L
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Obesity induced by other endocrinologic disorders (e.g., Cushing Syndrome)
* Current or history of treatment with medications that may cause significant weight gain for at least 3 months before this trial
* Current participation in an organized diet reduction program (or within the last 3 months)
* Currently using or have used within three months before this trial: pramlintide, sibutramine, orlistat, zonisamide, topiramate, phenteremine, or metformin
* Previous surgical treatment for obesity (excluding liposuction if performed more than one year before trial entry)
* History of major depressive disorder or a PHQ-9 (Patient Health Questionnaire-9) score of more than 15 within the last 2 years or history of other severe psychiatric disorders or diagnosis of an eating disorder
* Subjects with a lifetime history of a suicide attempt or history of any suicidal behavior within the past month before entry into the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2008-10-30 (Actual); Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (35):
- United States (25):
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Peoria, Arizona
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Endwell, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Norfolk, Virginia
- Canada (10):
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Mirabel, Quebec
  - Novo Nordisk Investigational Site, Sherbrooke, Quebec
  - Novo Nordisk Investigational Site, Trois-Rivières, Quebec
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Montreal

REFERENCES:
- [Result] O'Neil PM, Garvey WT, Gonzalez-Campoy JM, Mora P, Ortiz RV, Guerrero G, Claudius B, Pi-Sunyer X; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. EFFECTS OF LIRAGLUTIDE 3.0 MG ON WEIGHT AND RISK FACTORS IN HISPANIC VERSUS NON-HIPANIC POPULATIONS: SUBGROUP ANALYSIS FROM SCALE RANDOMIZED TRIALS. Endocr Pract. 2016 Nov;22(11):1277-1287. doi: 10.4158/EP151181.OR. Epub 2016 Aug 2. PMID 27482610
- [Result] Bays H, Pi-Sunyer X, Hemmingsson JU, Claudius B, Jensen CB, Van Gaal L. Liraglutide 3.0 mg for weight management: weight-loss dependent and independent effects. Curr Med Res Opin. 2017 Feb;33(2):225-229. doi: 10.1080/03007995.2016.1251892. Epub 2016 Nov 6. PMID 27817208
- [Result] Wadden TA, Hollander P, Klein S, Niswender K, Woo V, Hale PM, Aronne L; NN8022-1923 Investigators. Weight maintenance and additional weight loss with liraglutide after low-calorie-diet-induced weight loss: the SCALE Maintenance randomized study. Int J Obes (Lond). 2013 Nov;37(11):1443-51. doi: 10.1038/ijo.2013.120. Epub 2013 Jul 1. PMID 23812094
- [Result] McEvoy BW. Missing data in clinical trials for weight management. J Biopharm Stat. 2016;26(1):30-6. doi: 10.1080/10543406.2015.1094814. PMID 26418188
- [Result] Steinberg WM, Rosenstock J, Wadden TA, Donsmark M, Jensen CB, DeVries JH. Impact of Liraglutide on Amylase, Lipase, and Acute Pancreatitis in Participants With Overweight/Obesity and Normoglycemia, Prediabetes, or Type 2 Diabetes: Secondary Analyses of Pooled Data From the SCALE Clinical Development Program. Diabetes Care. 2017 Jul;40(7):839-848. doi: 10.2337/dc16-2684. Epub 2017 May 4. PMID 28473337
- [Result] O'Neil PM, Aroda VR, Astrup A, Kushner R, Lau DCW, Wadden TA, Brett J, Cancino AP, Wilding JPH; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Neuropsychiatric safety with liraglutide 3.0 mg for weight management: Results from randomized controlled phase 2 and 3a trials. Diabetes Obes Metab. 2017 Nov;19(11):1529-1536. doi: 10.1111/dom.12963. Epub 2017 Jul 21. PMID 28386912
- [Result] Davies MJ, Aronne LJ, Caterson ID, Thomsen AB, Jacobsen PB, Marso SP; Satiety and Clinical Adiposity - Liraglutide Evidence in individuals with and without diabetes (SCALE) study groups. Liraglutide and cardiovascular outcomes in adults with overweight or obesity: A post hoc analysis from SCALE randomized controlled trials. Diabetes Obes Metab. 2018 Mar;20(3):734-739. doi: 10.1111/dom.13125. Epub 2017 Nov 1. PMID 28950422
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 26 sites in the United States and 10 sites in Canada.
Pre-assignment Details: Subjects who lost at least 5% of screening body weight after 4 weeks and up to 12 weeks during the run-in were randomised in a 1:1 manner to receive either liraglutide 3.0 mg, or placebo for 56 weeks.
Period: Main Trial Period Through Week 56
Arm/Group | Lira 3.0 mg | Placebo
Started | 212 | 210
Completed | 159 | 146
Not Completed | 53 | 64
Not completed — Adverse Event | 18 | 18
Not completed — Lack of Efficacy | 0 | 2
Not completed — Protocol Violation | 8 | 5
Not completed — Withdrawal by Subject | 17 | 24
Not completed — Unclassified | 10 | 15
Period: Follow up Period (Week 56-68)
Arm/Group | Lira 3.0 mg | Placebo
Started | 159 | 146
Completed | 153 | 141
Not Completed | 6 | 5
Not completed — Protocol Violation | 1 | 1
Not completed — Unclassified | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 3.0 mg | Placebo | Total
Number analyzed (Participants) | 212 | 210 | 422
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.9) | 46.5 (11.0) | 46.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 165 | 343
  Male | 34 | 45 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 11 | 28
  Not Hispanic or Latino | 195 | 199 | 394
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 32 | 24 | 56
  White | 170 | 185 | 355
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 1 | 8
Co-morbidity status [Number; unit: participants] — Presence or absence of treated or untreated hypertension or dyslipidaemia
  participants
    Present | 94 | 96 | 190
    Absent | 118 | 114 | 232
Co-morbidity status and Body Mass Index (BMI) [Number; unit: participants] — Presence or absence of treated or untreated hypertension or dyslipidaemia
  participants
    Present and BMI (27-30) kg/m^2 | 3 | 6 | 9
    Present and BMI >=30 kg/m^2 | 91 | 90 | 181
    Absent and BMI >=30 kg/m^2 | 118 | 114 | 232
Smoking [Number; unit: participants]
  Yes | 20 | 22 | 42
  No | 192 | 188 | 380
Height [Mean (Standard Deviation); unit: meters] | 1.67 (0.09) | 1.67 (0.09) | 1.67 (0.09)
Weight at screening [Mean (Standard Deviation); unit: kg] | 106.7 (21.8) | 105.0 (22.4) | 105.9 (22.1)
Weight at randomisation [Mean (Standard Deviation); unit: kg] | 100.4 (20.8) | 98.7 (21.2) | 99.6 (21.0)
Body Mass Index (BMI) at screening [Mean (Standard Deviation); unit: kg/m^2] | 38.2 (6.2) | 37.5 (6.2) | 37.9 (6.2)
Body Mass Index (BMI) group (kg/m^2) at screening [Number; unit: participants]
  27-30 | 3 | 6 | 9
  30-35 | 69 | 80 | 149
  35-40 | 69 | 58 | 127
  Greater than or equal to 40 | 71 | 66 | 137
Body Mass Index (BMI) at randomisation [Mean (Standard Deviation); unit: kg/m^2] | 36.0 (5.9) | 35.2 (5.9) | 35.6 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change in Fasting Body Weight From Baseline
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: Last Observation Carried Forward, Full Analysis Set (includes all randomised subjects exposed to at least 1 dose of trial product and with at least 1 post-randomisation assessment of any efficacy endpoint.)
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
percentage | -6.11 (0.66) | -0.05 (0.63)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; The 3 co-primary endpoints (Outcome Measures 1, 2 and 3) were ranked (#1, 2, 3) and the hypotheses of equality between liraglutide and placebo for each were tested in a hierarchical manner; i.e. a conclusion of liraglutide superiority for a given co-primary endpoint could be drawn only if all preceding hypotheses of equality in the hierarchy had been rejected; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two sided, conducted at a 5% significance level; The analysis included treatment, gender, country and stratification factor(s) as fixed effects and randomisation value of the endpoint as covariate; Treatment Contrast = -6.06, 95% CI [-7.50 to -4.62]

2. Primary Outcome: Percentage of Subjects Who Maintained Their run-in Fasting Weight Loss From Week 0
Description: Subjects who had a weight regain less than or equal to 0.5% of weight from Week 0 were regarded as maintenance of run-in fasting weight loss. Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
percentage of subjects | 80.8 | 47.9
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Two sided, conducted at a 5% significance level; The analysis included treatment, gender, country, and stratification factor(s) as fixed effects and randomisation value of endpoint as covariate; Odds Ratio (OR) = 4.82, 95% CI [3.01 to 7.71]

3. Primary Outcome: Percentage of Subjects Who Lost More Than or Equal to 5% of Fasting Body Weight From Week 0
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
percentage of subjects | 50.5 | 21.9
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Two sided, conducted at a 5% significance level; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 3.86, 95% CI [2.44 to 6.09]

4. Secondary Outcome: Percentage of Subjects Who Lost More Than 10% of Fasting Body Weight From Week 0
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: Full Analysis Set (includes all randomised subjects exposed to at least 1 dose of trial product and with at least 1 post-randomisation assessment of any efficacy endpoint.)
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
percentage of subjects | 26.1 | 6.3
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Two sided, conducted at a 5% significance level; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 5.30, 95% CI [2.79 to 10.08]

5. Secondary Outcome: Percentage of Subjects With Weight Regain (Fasting) More Than or Equal to 5% From Week 0
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
percentage of subjects | 1.9 | 17.5
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Two sided, conducted at a 5% significance level; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 0.09, 95% CI [0.03 to 0.26]

6. Secondary Outcome: Percentage of Subjects With Weight Regain (Fasting) More Than or Equal to 10% From Week 0
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
percentage of subjects | 0 | 2.9

7. Secondary Outcome: Percentage of Subjects With Greater Than 50% of Fasting run-in Weight Loss Maintained From Week 0
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
percentage of subjects | 93.2 | 70.9
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Two sided, conducted at a 5% significance level; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 5.86, 95% CI [3.12 to 10.98]

8. Secondary Outcome: Percentage of Subjects With Greater Than 75% of Fasting run-in Weight Loss Maintained From Week 0
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
percentage of subjects | 87.4 | 54.4
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Two sided, conducted at a 5% significance level; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 6.02, 95% CI [3.65 to 9.92]

9. Secondary Outcome: Change From Baseline in Fasting Weight
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
kg | -5.7 (0.66) | 0.16 (0.63)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -5.86, 95% CI [-7.30 to -4.43]

10. Secondary Outcome: Change From Baseline in Fasting Weight for Subjects Completing the Main Trial Period and Entering the Follow-up Period
Description: Subjects were weighed having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 68
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 159 | 144
kg | -3.83 (0.82) | 0.41 (0.78)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -4.23, 95% CI [-6.04 to -2.43]

11. Secondary Outcome: Change From Baseline in Blood Pressure
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
mmHg
  Change in Systolic Blood Pressure | 1.31 (0.90) | 4.03 (0.87)
  Change in Diastolic Blood Pressure | 1.81 (0.64) | 2.15 (0.61)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Analysis is of treatment contrast, change in systolic blood pressure; Test type: Superiority or Other; p = 0.0068, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -2.72, 95% CI [-4.69 to -0.76]
Statistical Analysis 2: Comparison: Lira 3.0 mg vs Placebo; Analysis is of treatment contrast, change in diastolic blood pressure; Test type: Superiority or Other; p = 0.6386, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -0.34, 95% CI [-1.74 to 1.07]

12. Secondary Outcome: Change From Baseline in Pulse
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats/minute
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
beats/minute | 4.12 (0.68) | 3.15 (0.65)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.1968, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = 0.97, 95% CI [-0.51 to 2.45]

13. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Triglycerides
Description: Subjects were tested having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 187
mmol/L | 0.02 (0.04) | 0.12 (0.04)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0310, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -0.11, 95% CI [-0.20 to -0.01]

14. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Low Density Lipoprotein (LDL) Cholesterol
Description: Subjects were tested having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 187
mmol/L | 0.24 (0.05) | 0.33 (0.05)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.1098, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -0.09, 95% CI [-0.20 to 0.02]

15. Secondary Outcome: Change From Baseline in Fasting Lipid Profile: Total Cholesterol
Description: Subjects were tested having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 187
mmol/L | 0.22 (0.06) | 0.33 (0.06)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.1149, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -0.11, 95% CI [-0.24 to 0.03]

16. Secondary Outcome: Change From Baseline in Cardiovascular Biomarker: High Sensitivity C-reactive Protein (hsCRP)
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 185 | 174
nmol/L | -11.31 (4.62) | 1.70 (4.51)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0141, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -13.01, 95% CI [-23.40 to -2.64]

17. Secondary Outcome: Percentage of Subjects Meeting Metabolic Syndrome Criteria: ATP (Adult Treatment Panel) III at Week 56
Description: Metabolic syndrome status required at least 3 of 5 criteria met: Waist circumference (men ≥102cm, women ≥88cm); Triglycerides >1.7mmol/L; High density lipoprotein cholesterol (men <0.9mmol/L, women <1.1mmol/L) or on drug therapy; Blood pressure ≥130mmHg systolic or ≥85mmHg diastolic or on drug therapy; Fasting glucose ≥5.5mmol/L or on drug therapy.
Time Frame: Week 56
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
percentage of subjects | 31.4 | 36.7
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.1199, Regression, Logistic — Two sided, conducted at a 5% significance level; The analysis included treatment, gender, and stratification factor(s) as fixed effects and metabolic status and weight at baseline as covariates; Odds Ratio (OR) = 0.64, 95% CI [0.36 to 1.12]

18. Secondary Outcome: Change From Baseline in Waist Circumference
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
cm | -4.36 (0.62) | -0.86 (0.59)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -3.50, 95% CI [-4.84 to -2.15]

19. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg/m^2
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
kg/m^2 | -1.90 (0.22) | 0.15 (0.21)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -2.05, 95% CI [-2.53 to -1.57]

20. Secondary Outcome: Change From Baseline in Glycaemic Control Parameter: HOMA-B (Homeostasis Model Assessment - Beta Cell Function)
Description: Change in beta-cell function percent values from Week 0 (X%) to Week 56 (Y%) was calculated [X% - Y%]. Beta-cell function was derived from fasting plasma glucose readings in blood samples using the HOMA method, which is based on the assumption that normal-weight subjects without diabetes aged <35 years have median beta-cell function indexed at 100%.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 190 | 181
percent change | 8.51 (2.33) | 6.16 (2.27)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.3689, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = 2.35, 95% CI [-2.79 to 7.49]

21. Secondary Outcome: Change From Baseline in Glycaemic Control Parameter: HOMA-IR (Homeostasis Model Assessment - Insulin Resistance)
Description: Change in insulin resistance values from Week 0 (X) to Week 56 (Y) was calculated [X - Y]. Insulin resistance was derived from fasting serum insulin levels in blood samples using the HOMA method, which is based on the assumption that normal-weight subjects without diabetes aged <35 years have median insulin resistance indexed at 1.00.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: proportion
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 190 | 181
proportion | -0.01 (0.03) | 0.08 (0.03)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0053, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -0.10, 95% CI [-0.16 to -0.03]

22. Secondary Outcome: Change From Baseline in Glycaemic Control Parameter: Fasting Plasma Glucose (FPG)
Description: Subjects were tested having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
mmol/L | -0.52 (0.05) | -0.14 (0.05)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -0.38, 95% CI [-0.50 to -0.26]

23. Secondary Outcome: Change From Baseline in Glycaemic Control Parameter: Fasting Serum Insulin
Description: Subjects were tested having fasted (consumed only water) since midnight the night before the visit.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
pmol/L | 0.50 (0.67) | 2.35 (0.65)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p = 0.0147, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -1.85, 95% CI [-3.34 to -0.37]

24. Secondary Outcome: Change From Baseline in Glycaemic Control Parameter: HbA1c (Glycosylated Haemoglobin)
Description: Change in HbA1c percent values from Week 0 (X%) to Week 56 (Y%) was calculated [X% - Y%].
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage point
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 194 | 188
percentage point | -0.14 (0.03) | 0.13 (0.03)
Statistical Analysis 1: Comparison: Lira 3.0 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA — Two sided, conducted at a 5% significance level; [statistical method as in outcome 1, analysis 1]; Treatment Contrast = -0.27, 95% CI [-0.33 to -0.21]

25. Secondary Outcome: Number of Subjects Using Concomitant Medications (Antihypertensive Medications, Lipid Lowering Medications, or Antipsychotic Medications)
Description: Number of subjects using concomitant medications at Week 0 and Week 56, respectively
Time Frame: Week 0 and week 56
Population: as for outcome 4
Measure: Number; unit: Subjects
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
Subjects
  Antihypertensive drug - Week 0 | 65 | 66
  Antihypertensive drug - Week 56 | 63 | 63
  Antipsychotic drug - Week 0 | 18 | 25
  Antipsychotic drug - Week 56 | 20 | 29
  Lipid lowering drug - Week 0 | 45 | 45
  Lipid lowering drug - Week 56 | 52 | 50

26. Secondary Outcome: Binge Eating Scale Scores by Week and Severity
Description: Binge Eating Scale (BES) scores are based on responses to the Binge Eating Scale Questionnaire, a 16-item self-reporting diagnostic tool scaled 0-46 (Non-binging: 0-17; Moderate: 17-26; Severe: 27-46)
Time Frame: Week 0, week 50 and week 57
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Lira 3.0 mg | Placebo
Number analyzed (Participants) | 207 | 206
scores on a scale
  Week 0, baseline | 7.8 (5.6) | 7.8 (6.2)
  Week 50 | 6.6 (5.6) | 8.6 (7.0)
  Week 57 | 6.6 (5.8) | 6.9 (6.2)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were defined as occurring before randomisation and increasing in severity during treatment, or had onset on or after first day of randomised treatment and no later than 7 days after last day of randomised treatment.
Description: Safety analysis set were all randomised subjects who had been exposed to at least one dose of trial product.
Arm/Group | Lira 3.0 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 9/212 | 5/210
Other Adverse Events (participants affected / at risk) | 177/212 | 163/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 3.0 mg (N=212) | Placebo (N=210)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 3.0 mg (N=212) | Placebo (N=210)
Nasopharyngitis (Infections and infestations) | 36 (44) | 47 (63)
Sinusitis (Infections and infestations) | 16 (17) | 27 (33)
Upper Respiratory Tract Infection (Infections and infestations) | 26 (35) | 23 (33)
Influenza (Infections and infestations) | 15 (17) | 22 (25)
Urinary Tract Infection (Infections and infestations) | 15 (17) | 11 (11)
Bronchitis (Infections and infestations) | 7 (7) | 11 (15)
Nausea (Gastrointestinal disorders) | 101 (181) | 36 (55)
Constipation (Gastrointestinal disorders) | 57 (66) | 26 (28)
Diarrhoea (Gastrointestinal disorders) | 38 (53) | 26 (34)
Vomiting (Gastrointestinal disorders) | 35 (44) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 20 (25) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 14 (17) | 3 (4)
Abdominal Distension (Gastrointestinal disorders) | 13 (14) | 8 (9)
Eructation (Gastrointestinal disorders) | 11 (17) | 0 (0)
Flatulence (Gastrointestinal disorders) | 11 (17) | 8 (8)
Headache (Nervous system disorders) | 27 (42) | 26 (37)
Dizziness (Nervous system disorders) | 22 (35) | 18 (22)
Injection Site Haematoma (General disorders) | 17 (18) | 24 (32)
Fatigue (General disorders) | 17 (20) | 11 (12)
Injection Site Pain (General disorders) | 8 (9) | 11 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 20 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 13 (13)
Muscle Strain (Injury, poisoning and procedural complications) | 11 (13) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 11 (12)
Decreased Appetite (Metabolism and nutrition disorders) | 21 (22) | 3 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 11 (18) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones, e.g. a clinical trial report is available, including right to not release interim trial results, because this may lead to conclusions later shown to be incorrect. At trial end, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for a short time to protect intellectual property.